CLINICAL TRIAL: NCT01535183
Title: Irinotecan, Vincristine, Etoposide, Carboplatin, and Cyclophosphamide for Refractory or Relapsed Brain Tumor in Children and Adolescents
Brief Title: Irinotecan Combination Chemotherapy for Refractory or Relapsed Brain Tumor in Children and Adolescents
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-1201
Record Dates: First submitted 2012-02-07; First posted 2012-02-17 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Brain Tumor
Keywords: irinotecan; brain tumor; pediatrics; salvage therapy; chemotherapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan (Experimental)
  Interventions: Drug: Irinotecan combination chemotherapy

INTERVENTIONS:
Drug: Irinotecan combination chemotherapy — Irrinotecan 300㎎/㎡ d0 IVS mixed with D5W 500mL over 90min with atropine (-30 min)
  VCR 2㎎/㎡ d0 IV push
  Etoposide 100㎎/㎡ d0-d2 IV over 1hr
  Carboplatin 450㎎/㎡ d0 IV over 8hrs
  Cyclophosphamide 1,000㎎/㎡ d1 IVS with mesna
  Other Names: Camptosar (Pfizer) or Campto (Yakult Honsha)

SUMMARY:
The outcome of pediatric refractory or relapsed brain tumor is very dismal. Standard chemotherapy showed poor response to these patients. Although tandem high dose chemotherapy with hematopoietic progenitor stem cell rescues has been chosen as a potentially curative therapy for long term survival and better outcome is expected if tumor burden before transplantation reduced by chemotherapy, effective salvage chemotherapy for tumor reduction is not established yet. Irinotecan is a recently developed topoisomerase I inhibitor, and there are preclinical and phase I, II data which proved practical effects in brain tumors. In those studies, irinotecan was administered alone or in combination with one other drug.

Vincristine, etoposide, carboplatin, and cyclophosphamide have been used in many protocols for brain tumors but the result was very poor in refractory or relapsed cases. However, irinotecan can be effective with these multiple chemotherapeutic agents. According to the pilot study of irinotecan in combination with vincristine, etoposide, carboplatin and cyclophosphamide in the investigators center, 75% percent of total 12 patients reached more than stable disease, and 2 patients got long term complete remission only with this multi-agent combination chemotherapy. But the combination of irinotecan, vincristine, etoposide, carboplatin, and cyclophosphamide is not clinically studied yet especially for pediatric patients. To improve response rate and progression-free survival, the combination chemotherapy of irinotecan, vincristine, etoposide, carboplatin, and cyclophosphamide is designed for pediatric refractory or relapsed brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of brain tumor : embryonal brain tumor (medulloblastoma, CNS PNET, ATRT, etc), intracranial germ cell tumor
* Relapse or refractory state
* Prior therapy : Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. Patients are eligible 8 weeks from the day of stem cell infusion for autologous stem cell transplant, if hematological and all other eligibility criteria are met.
* Performance status: ECOG 0-2.
* Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

  1. Heart: a shortening fraction ≥ 28%
  2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal.
  3. Kidney: creatinine <2 × normal
* Patients must lack any active viral infections or active fungal infection.
* Patients (or one of parents if patients age < 20) should sign informed consent.

Exclusion Criteria:

* Pregnant or nursing women.
* Malignant (except brain tumor) or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
* Psychiatric disorder that would preclude compliance.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate response rate (more than stable disease) of combination chemotherapy | every 3 months
  - Response Criteria : WHO-based "Macdonald criteria", based on MRI
  1. Complete Response : disappearance of all enhancing tumor
  2. Partial Remission : more than 50 percentage decrease in the tumor measurement compared with the baseline scan
  3. Stable Disease : includes changes that do not meet criteria for CR, PR, or progressive disease (PD)
  4. Progressive Disease : more than 25 percentage increase in tumor measurement compared with the lesion size that defines the nadir, or smallest measurement, in the serial studies

SECONDARY OUTCOMES:
To evaluate adverse event | during chemotherapy and every follow up (3 times a week, up to 4 weeks)
  - Toxicity evaluation : CTC version 4.0. A copy of the current version of the CTCAE can be downloaded from the CTEP home page (http://ctep.info.nih.gov).
To evaluate progression-free survival | until last follow up (at least 1year)
  - Kaplan-Meier method will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, M.D., ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea